CLINICAL TRIAL: NCT02027753
Title: Efficacy and Safety of TrEating Type 2 Diabetic Patients With Inadequate Response to Metformin and DPP-4 Inhibitors by Adding Basal Insulin Therapy (Insulin Glargine)
Brief Title: Efficacy and Safety of Insulin Glargine in Patients With Type 2 Diabetes With Inadequate Control on DPP-4 Inhibitor Therapy
Acronym: TED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LANTUL06638; U1111-1149-1632 (Other: UTN)
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Metformin; Dipeptidyl-Peptidase IV Inhibitors; Sulfonylurea Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin glargine and Oral anti diabetic treatment(s) (Experimental): 1. Insulin glargine: Lantus
     * Add basal insulin: starting with 0.2 U/kg/day or 10 U/day
     * Adjust insulin glargine dose according to Fasting blood glucose
  2. Oral Anti Diabetic treatment(s): DPP-4 inhibitors and Metformin plus or minus Sulphonylurea - Only Sulphonylurea can either be omitted or reduced at the physician's discretion.
  Interventions: Drug: INSULIN GLARGINE; Drug: Metformin; Drug: DPP-4 inhibitor; Drug: Sulphonylurea

INTERVENTIONS:
Drug: INSULIN GLARGINE — Pharmaceutical form: solution Route of administration: subcutaneous
Drug: Metformin — Pharmaceutical form: tablet Route of administration: oral
Drug: DPP-4 inhibitor — Pharmaceutical form: tablet Route of administration: oral
Drug: Sulphonylurea — Pharmaceutical form: tablet Route of administration: oral

SUMMARY:
Primary Objective:

To investigate the efficacy(HbA1c) at 6 months after adding basal insulin therapy (insulin glargine) to dipeptidyl peptidase-IV (DPP-IV) and metformin plus or minus sulphonylurea

Secondary Objectives:

1. To assess the efficacy by adding insulin glargine
2. To assess insulin dose
3. Safety

DETAILED DESCRIPTION:
28 weeks (Screening: About 2 weeks/Treatment: 24 weeks (6 months)/Follow-up: 2 weeks)

ELIGIBILITY:
Inclusion criteria :

* Patients with type 2 Diabetes mellitus ≥ 20 aged
* Patients who are treated with DPP- 4 for at least 3 months before informed consent with metformin plus or minus sulphonylurea inadequately controlled with HbA1c ≥ 7.5%
* Be able and voluntarily agree to participate in this study by signing a written informed consent

Exclusion criteria:

* Diabetes patients other than Type 2 (eg. Type 1 Diabetes mellitus, pancreatic disease, secondary diabetes)
* HbA1c > 11% at screening
* History of continuous basal insulin treatment within 1 year before screening
* History of diabetic acidosis (including keto-acidosis) within 1 year before screening
* History of myocardial infarct, stroke or heart failure related admission within 3 months before screening
* History of drug or alcoholic abuse within 6 months before screening
* Weight change ≥ 5 kg within 3 months before screening
* History of hypoglycemic unawareness
* Systolic blood pressure >180 mmHg or diastolic blood pressure > 110 mmHg regardless of taking anti-hypertensive, or uncontrolled hypertension
* Active malignant cancer, major systemic disease, clinically significant diabetic retinopathy, macular edema necessitating laser treatment, abnormal clinical finding from physical examination, lab analysis, electrocardiogram or vital sign, which can be regarded as to prevent safe completion of clinical study or to make efficacy assessment difficult by investigator or co-investigator at screening
* Pregnant or lactating women
* Women of child bearing potential (Pre-menopause or not surgically infertile within 3 months before screening) who match two conditions below:
* Negative serum pregnancy test at screening
* Using medically proven effective contraceptive method
* Hypersensitivity to investigational drugs
* Lab finding at screening:
* Abnormal liver function: Alanine transaminase or Alkaline phosphatase > 3 times of upper limit of normal range
* Renal insufficiency: Men with serum Cr ≥ 1.5 mg/dL (≥ 133µmol/L), women with serum Cr ≥ 1.4 mg/dL (≥ 124 µmol/L)
* Use of anti-obese drug within 3 months before screening
* Has been using drugs that can influence glucose metabolism (systemic corticosteroid, thyroid hormone) within 3 months before screening or has possibility of using these drug during the investigational period
* Has participated in clinical studies of any investigational drugs within 3 months before screening
* Considered not physically or psychologically appropriate to participate in clinical study by investigator
* Not willing to comply with scheduled visit, self-inject insulin, or self-monitor blood glucose level

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Response rate (percentage of patients who meet the target HbA1c ≤7%) at week 24 (6 months) after adding insulin therapy | week 24 (6 months)

SECONDARY OUTCOMES:
Percentage of patients with HbA1c ≤7% | week 12 (3 months)
Change from baseline in HbA1c | week 12 (3 months), week 24 (6 months)
Percentage of patients with HbA1c ≤6.5% | week 12 (3 months), week 24 (6 months)
Change from baseline in Fasting Plasma glucose (FPG), 2hr-Postprandial Plasma Glucose | week 12 (3 months), week 24 (6 months)
Total daily insulin dose | week 24 (6 months)
Fasting blood glucose (FBG) values | During 3 consecutive days before baseline, week 12, Week 24
7-point Self Monitoring of Blood Glucose | During 2 days within 7 days before baseline, week 12, week 24
Weight change from baseline | week 24 (6 months)
Number of Patients with Hypoglycemic Events | up to 6 months
Number of Patients with Adverse Events | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Seoul, South Korea